CLINICAL TRIAL: NCT02300441
Title: HI-VISION - Hypotension Myocardial Ischemia-Vascular Events In Noncardiac Surgery Patients: a Cohort Evaluation: Pilot Study
Brief Title: HI-VISION Pilot Study
Acronym: HI-VISION
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: HI-VISION Pilot Study
Record Dates: First submitted 2014-10-20; First posted 2014-11-25 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2016-03

CONDITIONS: Postoperative Hypoxia
MeSH Terms: interventions — epicatechin gallate; Blood Pressure; Oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: ECG, blood pressure and oximetry

SUMMARY:
A prospective cohort pilot study of non-cardiac patients to determine the feasibility of recruiting 150 patients to undergo postoperative continuous hemodynamic monitoring for up to 3 days.

DETAILED DESCRIPTION:
Patient will start wearing the Philips' hemodynamic and ECG monitor in the Post Anaesthesia Care Unit (PACU). This device will continuously measure heart rate, pulse oxymetry, and ST-segments. The device will measure blood pressure every hour from 7 am to 10 pm and every 2 hours from 10 pm to 7 am.

Patients will have postoperative Troponin I monitoring and telephone follow-up at 30 days postop.

ELIGIBILITY:
Inclusion Criteria: We will enroll patients aged 45 years or older undergoing noncardiac surgery who fulfilled 2 or more of the following risk factors:

* History of coronary artery disease
* History of stroke or transient ischemic attack (TIA)
* History of hypertension
* History of diabetes
* History of peripheral vascular disease
* History of congestive heart failure
* Preoperative creatinine > 175 umol/L
* A planned admission for ≥48 hours
* Patients receiving a general or regional anesthetic

Exclusion Criteria:

* Patients unable to provide informed consent.
* Patients who undergo procedure performed under infiltrative or topical anesthesia.
* Patients previously enrolled in the HI-VISION Study.
* Patients who refuse 30-day follow-up.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 45 or greater who present for noncardiac surgery with 2 or more risk factors for heart disease and will be receiving a general or spinal anesthesia with an anticipated length of stay of 3 days or more.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Hypotension and Hypoxemia (baseline patterns and frequencies) | 10 months
  To identify baseline patterns and frequencies of hypotension and hypoxemia.

SECONDARY OUTCOMES:
Myocardial Ischemia (association between myocardial ischemia detected by the algorithm implemented by MX40 with Troponin I) | 10 months
  To determine the association between myocardial ischemia detected by the algorithm implemented by MX40 with Troponin I.
Myocardial Ischemia (delay in detecting myocardial ischemia based on MX40 monitoring versus Troponin I monitoring) | 10 months
  To determine the delay in detecting myocardial ischemia based on MX40 monitoring versus Troponin I monitoring.
Myocardial Ischemia (number of patients with missed clinically important hypotension, bradycardia, and hypoxia based on routine monitoring in clinical practice versus remote, automated, non-invasive hemodynamic monitoring) | 10 months
  To determine the number of patients with missed clinically important hypotension, bradycardia, and hypoxia based on routine monitoring in clinical practice versus remote, automated, non-invasive hemodynamic monitoring.
Myocardial Ischemia (delay in detecting clinically important hypotension, bradycardia, and hypoxia based on routine monitoring in clinical practice versus remote, automated, non-invasive hemodynamic monitoring.) | 10 months
  To determine the delay in detecting clinically important hypotension, bradycardia, and hypoxia based on routine monitoring in clinical practice versus remote, automated, non-invasive hemodynamic monitoring.

OTHER OUTCOMES:
Postoperative Pain (association between postoperative pain intensity and myocardial ischemia, nonfatal myocardial infarction, and cardiac mortality) | 10 months
  To determine the association between postoperative pain intensity and myocardial ischemia, nonfatal myocardial infarction, and cardiac mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Philip J. Devereaux, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Juravinski Hospital, Hamilton, Ontario, Canada